CLINICAL TRIAL: NCT01247766
Title: Post-marketing Observational Study Assessing the Long-term Safety of Abatacept Using a Population-based Cohort of Rheumatoid Arthritis Patients in the Province of British Columbia
Brief Title: Safety Study of Abatacept to Treat Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Arthritis Research Centre of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: IM101-213
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with rheumatoid arthritis (RA) who receive abatacept
- Patients with RA who receive BDM drugs: biologic disease-modifying (BDM)
- Patients with RA who receive non-biologic DMARDs: disease-modifying anti-rheumatic drugs (DMARDs)

SUMMARY:
The purpose of this study is to compare the incidence rates of infection, malignancy and death among patients with rheumatoid arthritis who are treated with abatacept and those who are treated with other anti-rheumatic medications for rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis
* Receipt of abatacept, other biologic disease-modifying drug, or any non- biologic disease-modifying anti-rheumatic drug
* Age 18 years or older

Exclusion Criteria:

* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of British Columbia who have received health care service for rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 6367 (Actual)
Dates: Start 2010-12-31 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Serious infection | Every 2 years throughout the study
Incidence rates of malignancy | Every 2 years throughout the study
  (total, lymphoma, lung cancer, breast cancer, colorectal cancer)
Total mortality | Every 2 years throughout the study

SECONDARY OUTCOMES:
Multiple sclerosis | Every 2 years throughout the study
  To determine the incidence rate of multiple sclerosis (MS) in RA patients treated with abatacept and to compare this rate with the rate in RA patients matched for age, gender, RA duration and DMARD use, after adjusting for other potential confounders.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm